CLINICAL TRIAL: NCT02890654
Title: Idiopathic Scoliosis Surgery in Adolescents ; Earnings a Multidisciplinary Management of Pain and Quality of Life
Brief Title: Scoliosis and Quality of Life of Adolescents
Acronym: SQUAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31-15-7475
Record Dates: First submitted 2016-07-06; First posted 2016-09-07 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Scoliosis
Keywords: Teenagers; Multidisciplinary approach; Pain; Surgery
MeSH Terms: conditions — Scoliosis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Teenagers with scoliosis: Patients will be evaluated at three times during the study :
  * First time measure : 1 month before the scoliosis surgery
  * Second time measure : 3 months after the scoliosis surgery
  * Third time measure : 1 year after the scoliosis surgery
  Interventions: Other: First time measure; Other: Second time measure; Other: Third time measure

INTERVENTIONS:
Other: First time measure — * Initial Interview
  * Initial Survey,
  * Quality of life Scale
  * Kinesitherapy Review
  * Anxiety Scale
Other: Second time measure — * Kinesitherapy review
  * Second survey including numeric scale of pain
  * Anxiety scale
  * Scoliosis Research Society 22 quality of life scale
Other: Third time measure — * Scoliosis Research Society 22 quality of life Scale
  * Anxiety scale
  * Numeric scale of pain
  * Kinesitherapy review

SUMMARY:
Around the scoliosis surgery, the pain (pre or post operative, physical, psychological, fantasy or real) is a major concern for adolescents and their families. She is also a key concern of caregivers, both its assessment and management is complex. this pain involved predominantly in the quality of life of these teenagers today who will become the adults of tomorrow.

To date in France, no study aims to describe and evaluate the effect of a multidisciplinary approach and its impact on the quality of life of these young people made.

The present study wish to prevent, anticipate and limit the short, medium and long-term morbidity. Focus will be on pain and its management, on preparing for surgery, hospitalization, follow-up after surgery, rehabilitation until recovery.

Help teens reclaim their bodies after the changes caused by the intervention is a major issue.

This study believe that support good quality, adapted to patient needs will limit operating and postoperative pain in the medium and long term.

Medical team developed special attention around the teenagers that are operated for scoliosis (teen groups and parent groups, interview before the operation and counseling, physiotherapy support ...).

The present study would systematize data collections in order to have a comprehensive and accurate assessment of the care.

The qualitative research will focus on the multidisciplinary care in an effort to evaluate the whole course of these teenagers, their experience and to identify efforts to put in place to optimize the current care.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed for idiopathic scoliosis with indication for surgery
* Patients monitored and operated at the Children Hospital of Toulouse

Exclusion Criteria:

* Opposition to the participation
* Spine deformations other than scoliosis
* Non idiopathic scoliosis

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Teenagers with diagnosis of idiopathic scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Comparison of quality of life before and after the surgery with Scoliosis Research Society 22 questionary | 1 Month before surgery
Comparison of quality of life before and after the surgery with Scoliosis Research Society 22 questionary | 3 Month after surgery
Comparison of quality of life before and after the surgery with Scoliosis Research Society 22 questionary | 6 months after the surgery

SECONDARY OUTCOMES:
Comparison of pain before and after the surgery as assessed by visual scale of pain | 1 Month before surgery, 3 months and 6 months after the surgery
Comparison of pain before and after the surgery as assessed by visual scale of pain | 1 Month before surgery
Comparison of pain before and after the surgery as assessed by visual scale of pain | 3 Months after surgery
Comparison of anxiety before and after the surgery as assessed by anxiety scale | 6 months after the surgery
Patient global satisfaction before and after the surgery as assessed by oriented interviews | 1 Month before surgery
Patient global satisfaction before and after the surgery as assessed by oriented interviews | 6 months after surgery
Evaluation of scoliosis typography with kinesitherapy complete assessment using radiography of the back | 1 Month before surgery
Evaluation of scoliosis typography with kinesitherapy complete assessment using radiography of the back | 3 months after the surgery
Evaluation of scoliosis typography with kinesitherapy complete assessment using radiography of the back | 6 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Agnès SUC, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- Children Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided